CLINICAL TRIAL: NCT02779920
Title: Feasibility of Endoscopic Pylorotomy in the Treatment of Refractory Gastroparesis, Pilot Study.
Acronym: GASTROPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I15002 (GASTROPOP)
Record Dates: First submitted 2016-02-23; First posted 2016-05-23 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Gastroparesis
Keywords: refractory gastroparesis; per oral pyloromyotomy
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Per oral pylorotomy (Experimental): Patients with gastroparesis (significant prolongation of gastric emptying) not improved prokinetic and antiemetic treatments undergoing per oral pylorotomy
  Interventions: Procedure: per oral pylorotomy

INTERVENTIONS:
Procedure: per oral pylorotomy — The procedure is endoscopic pylorotomy. The standard procedure consists in the realization of a longitudinal incision of 2 cm at the anterior surface of the gastric antrum at 5 cm from the pylorus after a submucosal injection of a solution containing 85% saline 10% glycerol and 5% fructose. This longitudinal incision serve as an input for producing a submucosal tunnel dissected fibers gastric submucosa step. The internal circular of the pyloric muscle is then severed fiber after fiber over its entire length and its entire thickness. Once the pyloric section completed, the tunnel inlet will be closed by means of hemostatic clips.

SUMMARY:
Gastroparesis is a common chronic condition, disabling the limited therapeutic resources justifying the exploration of new therapeutic possibilities.

By analogy to the technique of Per Oral Endoscopic Myotomy (POEM), we believe that myotomy pyloric muscle (POP = Per Oral Pyloromyotomy) endoscopically could become a treatment of choice in the refractory gastroparesis with drug treatments by attacking the pyloric obstacle often spastic that counteracts an effective gastric emptying.

DETAILED DESCRIPTION:
Experimental study, prospective, single-center, POP feasibility pilot in the treatment of refractory gastroparesis.

Patients with gastroparesis (significant prolongation of gastric emptying) unimproved by prokinetic treatment and meet all the eligibility criteria will be included after a period of reflection of two weeks minimum.

20 patients will be prospectively included 10 patients with diabetic gastroparesis, 10 patients with non-diabetic gastroparesis (post-surgical, post-Sjogren, idiopathic).

POP will be performed under general anesthesia in intubated-ventilated patients using a carbon dioxide (CO2) inflator. The published standard technique and learned by our team on the pig model will be conducted: submucosal tunnel at the anterior surface of the gastric antrum starting 3-5 cm proximal to the pylorus front section to the fiber by fiber to the muscular pyloric, then closing the inlet tunnel by hemostatic clips.

An evaluation of symptoms by the Gastroparesis Cardinal Symptom Index (ISCC) of the quality of life of the patient Assessment of upper gastrointestinal disorders-Quality Of Life (PAGI-QoL), SF-36 and gastrointestinal Quality of Life Index (GIQLI ) and gastric emptying by a scintigraphic gastric emptying will be carried out at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient with refractory gastroparesis to drug treatment (post-diabetic, post-Sjogren, postsurgical or idiopathic)
* Signed Consent
* Affiliate or beneficiary of a French social security scheme

Exclusion Criteria:

* Contraindications to gastroesophageal gastroduodenal endoscopy,
* Early Unable to follow protocol,
* Contraindications to general anesthesia,
* Can not Stop anticoagulants for the gesture,
* Can not stop antiplatelet agents for the gesture,
* Pregnant or lactating women,
* Gastric resection surgery History of pyloric
* Patients under guardianship, curatorship or safeguard justice,
* Disorders of hemostasis against-indicating the endoscopic procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of technical success for endoscopic pylorotomy on the total number of gestures. | 3 months
  Technical feasibility will be the feasibility of endoscopic pylorotomy gesture by the technique of the tunnel.

SECONDARY OUTCOMES:
Incidence of adverse events of pylorotomy | 3 months
  analysis of adverse events during the 3 months following the pylorotomy (including perforation per-gesture, bleeding post-gesture)
Ratio between the diameter of the pyloric canal and the pyloric pressure | Baseline and 3 months
  Evaluation of the pyloric compliance by the Endolumenal Functional Lumen Imaging Probe (EndoFLIP) system before the procedure and at 3 months, depending on etiology.
Assessment of gastric emptying scintigraphy | baseline and 3 months
  Assessment of gastric emptying scintigraphy before the procedure and at 3 months by measuring the half gastric emptying time and percentage retention to 4 hours
Assessment of gastroparesis severity symptom using the Gastroparesis Cardinal Symptom Index (GCSI) | Baseline, 1 month and 3 month
  Evaluation of the severity of gastroparesis symptom using the GCSI questionnaire
Assessment of Quality of Life in Upper Gastrointestinal Disorders (PAGI-QOL) | Baseline, 1 month and 3 month
  Evaluation of the quality of life of patient with Upper Gastrointestinal Disorders using PAGI-QOL questionnaire
Assessment of Quality of Life in Gastrointestinal disease (GIQLI) | Baseline, 1 month and 3 month
  Evaluation of quality of life of patients with gastrointestinal Disease using GIQLI questionnaire
Assessment of functional health and well-being from the patient's point of view (SF-36) | Baseline, 1 month and 3 month
  Evaluation of of functional health and well-being from the patient's point of view using SF-36 questionnaire
Consumption of gastric prokinetic drugs | 3 months
  Data collecting about domperidone, metoclopramide and erythromycin consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie Jacques, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- CHU de LIMOGES, Limoges, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jacques J, Pagnon L, Hure F, Legros R, Crepin S, Fauchais AL, Palat S, Ducrotte P, Marin B, Fontaine S, Boubaddi NE, Clement MP, Sautereau D, Loustaud-Ratti V, Gourcerol G, Monteil J. Peroral endoscopic pyloromyotomy is efficacious and safe for refractory gastroparesis: prospective trial with assessment of pyloric function. Endoscopy. 2019 Jan;51(1):40-49. doi: 10.1055/a-0628-6639. Epub 2018 Jun 12. PMID 29895073